CLINICAL TRIAL: NCT04691713
Title: CD276 CAR-T for Patients With Advanced CD276+ Solid Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: PersonGen BioTherapeutics (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PG-CART-276-001
Record Dates: First submitted 2020-12-07; First posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: CAR; Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Targeting CD276 autologous chimeric antigen receptor T cells (Experimental)
  Interventions: Drug: Targeting CD276 autologous chimeric antigen receptor T cells

INTERVENTIONS:
Drug: Targeting CD276 autologous chimeric antigen receptor T cells — Chimeric antigen receptor T cells (car-t) is one of the most effective therapies for malignant tumors (especially hematological tumors). Like other immunotherapies, the basic principle is to use the patient's own immune cells to clear cancer cells. Chimeric antigen receptor (car) is the core component of car-t, which endows T cells with the ability to recognize tumor antigens in an independent manner, which enables car modified T cells to recognize a wider range of targets than natural T cell surface receptors (TCR). The basic design of car includes a tumor associated antigen binding region (usually derived from scFv segment of monoclonal antibody antigen binding region), transmembrane region and intracellular signal region. The selection of target antigen is a key determinant for the specificity and effectiveness of car and the safety of genetically modified T cells.

SUMMARY:
This study is a clinical study of CD276 CAR-T in the treatment of patients with advanced solid tumors. The purpose is to evaluate the safety and effectiveness of targeting CD276 auto-chimeric antigen receptor T cells in the treatment of CD276-positive advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Age 3-70
* Expected survival time ≥ 12weeks
* ECOG 0-2
* At least second-line or above chemotherapy failed
* According to the evaluation criteria for the efficacy of solid tumors (RECIST 1.1), at least one measurable lesion (non-nodular lesion with longest diameter ≥10mm, or nodular lesion with short diameter ≥15mm)
* Liver and kidney function, heart and lung function meet the following requirements:

  1. Creatinine is within the normal range;
  2. Left ventricular ejection fraction ≥ 45%;
  3. Baseline blood oxygen saturation>91%;
  4. Total bilirubin≤1.5×ULN; ALT and AST≤2.5×ULN
* Understand the trial and have signed the informed consent

Exclusion Criteria:

* Those who have graft-versus-host disease (GVHD) or need to use immunosuppressive agents
* Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive and peripheral blood HBV DNA titer test is not within the normal reference range; hepatitis C virus (HCV) antibody positive and peripheral blood HCV RNA positive; human immunodeficiency virus (HIV) Antibody positive; CMV DNA test positive; Syphilis test positive
* Severe heart disease
* Systemic diseases judged by the investigator to be unstable: including but not limited to severe liver, kidney or metabolic diseases that require medication
* Within 7 days before screening, there are active infections or uncontrollable infections that require systemic treatment (except for mild urogenital infections and upper respiratory tract infections)
* Women who are pregnant or breastfeeding, and female subjects who plan to become pregnant within 1 year after cell reinfusion, or male subjects whose partners plan to become pregnant within 1 year after cell reinfusion
* Those who have received CAR-T therapy or other genetically modified cell therapy before screening
* Subjects who are receiving systemic steroid therapy at the time of screening and the investigator determines that they need long-term systemic steroid therapy during the treatment period (except for inhaled or topical use)
* Participated in other clinical studies within 3 months before screening
* Central nervous system metastases are known to occur and for suspected central nervous system metastases, head MRI examination is required to rule out
* Patients with partial or complete intestinal obstruction and complete biliary obstruction that cannot be relieved by active treatment
* With more than a moderate amount of ascites, or after conservative medical treatment (such as diuresis, sodium restriction, excluding ascites drainage) for 2 weeks, the ascites still shows a progressive increase
* According to the researcher's judgment, it does not meet the situation of cell preparation
* Situations that other researchers think are not suitable for inclusion

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-02-26 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
ORR 3 | Three months after CAR T cell infusion
  3-month objective response rate

CONTACTS AND LOCATIONS:
Locations (1):
- Bin Hu Hospital, Hefei, Anhui, China